CLINICAL TRIAL: NCT06391645
Title: Nerve Growth Factor Encapsulated With 2-methacryloyloxyethyl Phosphorylcholine Nanocapsules in the Treatment of Amyotrophic Lateral Sclerosis
Acronym: NATURAL
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing University of Chemical Technology (Unknown); Beijing Healthunion Cardio-Cerebrovascular Disease Prevention and Treatment Foundation (Unknown)
Responsible Party: Principal Investigator, yilong Wang, Executive Vice-President, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HX-A-2023027
Record Dates: First submitted 2024-03-08; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: nerve growth factor; amyotrophic lateral sclerosis; 2-methacryloyloxyethyl phosphorylcholine
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Hereditary Sensory and Autonomic Neuropathies | interventions — Nerve Growth Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MPC-NGF T1 (Experimental): 19.2mg MPC wrapped NGF per week for 13 times
  Interventions: Drug: Nerve Growth Factor
- MPC-NGF T2 (Experimental): 11.84mg MPC wrapped NGF per week for 13 times
  Interventions: Drug: Nerve Growth Factor
- X-NGF (Active Comparator): 19.2mg NGF per week for 13 times
  Interventions: Drug: Nerve Growth Factor

INTERVENTIONS:
Drug: Nerve Growth Factor — intravenously injection

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is one of the most lethal neurodegenerative diseases, with most patients dying from respiratory failure 3-5 years after the onset. The purpose of this study is to explore the efficacy and safety of nerve growth factor (NGF) encapsulated with 2-methacryloyloxyethyl phosphorylcholine (MPC) nanocapsules in the treatment of ALS patients.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is one of the most lethal neurodegenerative diseases. Most patients die due to respiratory failure 3-5 years after disease onset. Due to the low permeability and blocking of the blood-brain barrier (BBB) on more than 95% of all kinds of drugs, the drug treatment of ALS is relatively limited. Although a series of studies have been carried out on new therapies to ALS, such as monoclonal antibodies represented by ozanezumab and antisense oligonucleotides represented by tofersen, the conclusions are mostly limited to safety evaluation.

Nerve growth factor (NGF) provides protection and/or regeneration for neurons in the peripheral and central nervous system (CNS), which is considered to be a nerve regeneration agent with great therapeutic potential. The phase I clinical trial of intravenous recombinant human nerve growth factor (rhNGF) showed that, on the premise of ensuring safety, only a trace of NGF (3.6-7.38 ng/ml within 5 minutes) was detected in the plasma samples of the subjects who were injected with rhNGF 1.0 μg/kg (the maximum dose of this trial design).

In purpose of improving the therapeutic effect of NGF, the investigators plan to encapsulate NGF in nanoparticles linked by 2-methacryloyloxyethyl phosphorylcholine (MPC), consisting of one molecule of choline and one molecule of acetylcholine analog. After intravenous administration, the drug particles are effectively delivered to the CNS via receptor-mediated transcytosis (RMT) with the help of acetylcholine transporter and choline transporter widely expressed on brain capillary endothelial cells. The animal experiments have confirmed that intravenous injection of MPC encapsulated NGF capsule [n(NGF)] can effectively prolong the survival time of SOD1G93A mice, reduce the body weight loss and delay the time of dyskinesia onset compared with NGF. Similar results were obtained in the rhesus monkey model.

The purpose of this study is to explore the efficacy and safety of NGF encapsulated with MPC nanocapsules in the treatment of ALS patients.

This is a prospective, randomized, open-label, blinded endpoint (PROBE) clinical trial. The trial planned to enroll 60 ALS patients, aged 18-80 years, with disease duration 6 months to 3 years, with forced vital capacity (FVC) ≥ 85% of predicted value.

Patients will be randomly assigned to one of the following 3 groups at 1:1 ratio.

Treatment group 1: NGF 60ml wrapped in MPC nanomaterials (dose was given as 320 μg/ml) was injected intravenously every week for 12 weeks, including one administration at the starting point for a total of 13 times, as well as maintaining original basic drugs and rehabilitation treatment.

Treatment group 2: NGF 37ml wrapped in MPC nanomaterials (dose was given as 320 μg/ml) was injected intravenously every week for 12 weeks, including one administration at the starting point for a total of 13 times, as well as maintaining original basic drugs and rehabilitation treatment.

Control group: NGF 60ml (dose was given as 320 μg/ml) was injected intravenously every week for 12 weeks, including one administration at the starting point for a total of 13 times, as well as maintaining original basic drugs and rehabilitation treatment.

Face to face interviews will be made on baseline, 28±4 days after randomization, 84±7 days after randomization and 120±7 days after randomization. Online interviews will be made on 180±14 days and 1 year ±14 days after randomization.

The primary outcome, Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) scores of ALS patients in the treatment group and the control group after 3 months of NGF injection, will be compared by Wilcoxon rank sum test, and β and 95% confidence interval (CI) will be calculated. The survival / mortality of ALS patients in treatment group and control group will be analyzed by COX regression model, and hazard ratio (HR) value and 95%CI were be calculated. Survival curve will be calculated by Nelson-Aalen cumulative risk curve, and Gray's test will be used for comparison between groups.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old;
2. Confirmed or possible familial or sporadic ALS diagnosed according to the revised El Escorial criteria;
3. 6 months ≤disease duration ≤ 3 years, (onset time is defined as the time of the first occurrence of myasthenia);
4. Forced vital capacity (FVC) ≥ 85% of predicted value (based on gender, height and age);
5. Informed consent signed.

Exclusion Criteria:

1. Patients undergoing endotracheal intubation, non-invasive or mechanical ventilation;
2. Patients with diaphragmatic pacemakers;
3. Allergy to any component of the investigational medication, or any other allergic history that researchers deem necessary to be vigilant about;
4. Local skin infection or other suspicious signs of infection at the injection site;
5. Known hemorrhagic tendency (including but not limited to: platelet count <100×109/ L; on therapy of heparin, activated partial thromboplastin time (APTT) ≥35s; on therapy of warfarin, international normalized ratio (INR) >1.7; on therapy of novel oral anticoagulants; with direct thrombin or factor Xa inhibitor; accompanied with coagulopathy such as hemophilia);
6. Severe cardiac insufficiency before randomization (comply with New York College of Cardiology (NYHA) Cardiac Function Class III, IV);
7. Suffering from infectious diseases: hepatitis, tuberculosis, acquired immunodeficiency syndrome, etc;
8. Psychiatric disorders diagnosed according to Diagnostic and Statistical Manual of Mental Disorders (DSM-V) diagnostic criteria; or with suicidal intentions;
9. Women/men with desire to conceive during the experiment, and patients with pregnancy and lactation;
10. Difficulty in verbal communication, inability to communicate, understand or follow instructions, inability to cooperate with treatment and evaluation;
11. Combining with history of alcohol and drug abuse;
12. Unable to cooperate in follow-up due to geographical or other reasons;
13. Patients participated in other clinical trials or used other biologics, drugs, or devices under study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) | 84±7 days
  Change in Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) score (ALSFRS-R scores from 0 to 48, score decline indicates worse outcome of ALS patients, or disease progression and disability).

SECONDARY OUTCOMES:
Endpoint events | 28±4 days, 84±7 days, 120±7 days, 180±14 days, 1 year ±14 days
  The incidence of endpoint events (survival/mortality, tracheotomy/permanent respiratory, gastrostomy) of ALS patients.
Tolerance | 28±4 days, 84±7 days
  Tolerance of ALS patients during treatment: defined as percentage of subjects able to continue the investigational drug until planned discontinuation
Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) | 28±4 days, 120±7 days, 180±14 days, 1 year ±14 days
  Change in Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) score (ALSFRS-R scores from 0 to 48, score decline indicates worse outcome of ALS patients, or disease progression and disability).
Lung function: forced vital capacity | 28±4 days, 84±7 days, 120±7 days
  Forced vital capacity in millilitre of ALS patients. Value decline indicates worse outcome of ALS patients, or disease progression and disability.
Lung function: slow vital capacity | 28±4 days, 84±7 days, 120±7 days
  Slow vital capacity in millilitre of ALS patients. Value decline indicates worse outcome of ALS patients, or disease progression and disability.
Lung function: transcutaneous oxygen saturation | 28±4 days, 84±7 days, 120±7 days
  Transcutaneous oxygen saturation in % of ALS patients. Value decline indicates worse outcome of ALS patients, or disease progression and disability.
Muscle involvement | 120±7 days
  Muscle involvement will be assessed by needle electromyography, which analyzes muscle damage qualitatively based on spontaneous, motor unit action potential and recruitment. More muscle involvement indicates worse outcome of ALS patients, or disease progression and disability.

OTHER OUTCOMES:
Medullary function | 28±4 days, 84±7 days, 120±7 days
  Change in Center for Neurologic Study Bulbar Function Scale (CNS-BFS) score (from 21 to 105, score increase indicates worse outcome of ALS patients, or disease progression and disability).
Cognitive function | 120±7 days
  Change in Edinburgh Cognitive and Behavioural ALS Screen (ECAS) score (from 0 to 136, score decline indicates worse outcome of ALS patients, or disease progression and disability).
Wexner continence grading scale | 84±7 days, 120±7 days
  Change in Wexner continence grading scale score (from 0 to 30, score increase indicates worse outcome of ALS patients, or disease progression and disability).
Overactive Bladder Syndrome Score (OABSS) | 84±7 days, 120±7 days
  Change in Overactive Bladder Syndrome Score (OABSS, from 0 to 15, score increase indicates worse outcome of ALS patients, or disease progression and disability).
Amyotrophic Lateral Sclerosis Assessment Questionnaire-40 (ALSAQ-40) | 84±7 days, 120±7 days
  Change in Amyotrophic Lateral Sclerosis Assessment Questionnaire-40 (ALSAQ-40) score (from 40 to 200, score decline indicates worse outcome of ALS patients, or disease progression and disability).
Motor unit count | 28±4 days, 84±7 days
  Motor unit count analyzes muscle damage quantitatively based on motor unit number index (MUNIX) and motor unit size index (MUSIX). Value decline indicates worse outcome of ALS patients, or disease progression and disability.
Amplitude of Compound Muscle Action Potential (CMAP) | 28±4 days, 84±7 days
  Amplitude of Compound Muscle Action Potential (CMAP) analyzes muscle damage quantitatively. Value decline indicates worse outcome of ALS patients, or disease progression and disability.
Neurofilament light chain (NFL) | 28±4 days, 84±7 days
  The level of neurofilament light chain (NFL) in blood of ALS patients. Value increase indicates neuroinflammation or nerve damage.
Cystatin C | 28±4 days, 84±7 days
  The level of cystatin C in blood of ALS patients. Value increase indicates neuroinflammation or nerve damage.
Rasch Overall ALS Disability Scale (ROADS) | 28±4 days, 84±7 days, 120±7 days
  Change in Rasch Overall ALS Disability Scale (ROADS) score (from 0 to 56, score decline indicates worse outcome of ALS patients, or disease progression and disability).
Safety outcomes: incidence of adverse events | 28±4 days, 84±7 days
  Incidence of adverse events of ALS patients 28±4 days, 84±7 days after treatment: containing headache, Visual Analogue Scale (VAS), Brief Pain Inventory (BPI -9), local injection stimulation and local infection.
Safety test: blood routine | 28±4 days, 84±7 days, 120±7 days
  To collect blood samples and test for blood routine of ALS patients. Common laboratory abnormalities including hemoglobin<115g/l, or neutropenia<1.8*10^9/l, etc.
Safety test: liver function | 28±4 days, 84±7 days, 120±7 days
  To collect blood samples and test for liver function of ALS patients. Common laboratory abnormalities including glutamic pyruvic transaminase>41.0U/l, or glutamic oxaloacetic transaminase>42.0U/l, etc.
Safety test: renal function | 28±4 days, 84±7 days, 120±7 days
  To collect blood samples and test for renal function of ALS patients. Common laboratory abnormalities including creatinine>93.3μmol/l, with or without estimated glomerular filtration rate<90ml/min, etc.
Safety test: blood coagulation function | 28±4 days, 84±7 days, 120±7 days
  To collect blood samples and test for blood coagulation function of ALS patients. Common laboratory abnormalities including d-dimer>1.5μg/ml, or activated partial thromboplastin time>36.5seconds, etc.
Safety test: urine routine | 28±4 days, 84±7 days, 120±7 days
  To collect urine samples and test for urine routine of ALS patients. Common laboratory abnormalities including positive urine occult blood, or positive urine leucocyte etc.
Safety test: 12-lead electrocardiogram | 28±4 days, 84±7 days, 120±7 days
  To collect 12-lead electrocardiogram of ALS patients. Common abnormalities including ST segment elevation, or prolonged PR interval, or prolonged QT interval, etc.
Safety outcomes: adverse events (AE) and severe adverse events (SAE) | 28±4 days, 84±7 days, 120±7 days, 180±14 days, 1 year ±14 days
  Adverse events (AE) and severe adverse events (SAE): all AE and SAE in the trial will be recorded in the case report form.

IPD SHARING:
Plan to Share IPD: No